CLINICAL TRIAL: NCT04538443
Title: Impact of Chronic Kidney Disease on Children Functional Capacity and Their Families' Quality of Life: A Cross Sectional Study
Brief Title: Impact of CKD on Children and Their Families
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaymaa Rushdy Mahmoud, principal investigator, Cairo University
Other Study IDs: CKD comorbidity
Record Dates: First submitted 2020-08-30; First posted 2020-09-04 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D
Keywords: CKD; hemodialysis; functional capacity; QoL
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Functional Residual Capacity; Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hemodialysis group: One hundred children with ESRD who are treated with hemodialysis and their caregivers will participate in this study. They will be recruited from Nephrology Unit at Abo-Elreesh Hospital, Cairo University
  Interventions: Other: functional capacity; Other: muscle strength; Other: Quality of life of children; Other: Quality of life of families

INTERVENTIONS:
Other: functional capacity — impact of hemodialysis on functional capacity in children with CKD
Other: muscle strength — impact of hemodialysis on muscle strength in children with CKD
Other: Quality of life of children — impact of hemodialysis on Quality of life in children with CKD
Other: Quality of life of families — impact of hemodialysis on Quality of life of families of children with CKD

SUMMARY:
Based on the available literatures, previous studies have investigated the impact of CKD and dialysis on patient's health among adult and elderly population. As far as we know, this is the first empirical study that investigates the impact of CKD on children functional capacity and their families QOL.

DETAILED DESCRIPTION:
The current study will be done to investigate the long term effect of the CKD itself on different dimensions of the child health to understand the unique characteristics of pediatric CKD. Also, it will be beneficial for designing a comprehensive physical therapy protocol for prevention of different complications and to improve their wellbeing healthcare. Additionally, it will be beneficial to determine the family and parental stresses and to build the rehabilitation plan for the child considering the possible family issues regarding the child condition.

ELIGIBILITY:
Inclusion Criteria:

* Age from eight to twelve years.
* Both genders.
* Diagnosed with ESRD (stage 5) based on the glomerular filtration rate (GFR < 15 mL/minute/1.73 m2).
* Able to understand and follow instructions during assessment procedures.
* Willing to participate in the study and attend the assessment procedures.

Exclusion Criteria:

Children of the following criteria will be excluded from the study:

* Cardiopulmonary disorders
* Uncontrolled hypertension
* Unstable angina
* Severe uncontrolled diabetes
* Neurological or cognitive disorders with functional deficits
* Significant cerebral or peripheral vascular disease.

Ages: 8 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: One hundred children with ESRD who are treated with hemodialysis and their caregivers will participate in this study. They will be recruited from Nephrology Unit at Abo-Elreesh Hospital, Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
functional capacity | 6 months
  6 minute walking test is commonly used to evaluate functional capacity in children with CKD. It is a simple, practical, reliable, and valid measure of submaximal exercise capacity in healthy children and children with chronic disease or neuromuscular disorders or cardiopulmonary disease

SECONDARY OUTCOMES:
muscle strength | 6 months
  Hand grip strength HGS is a noninvasive and reliable method for assessment of muscle power and nutritional status in CKD children
quality of life of children | 6 months
  The Arabic version of the PedsQLTM 4.0 Generic Core Scales version proved to be understandable and feasible to use. It showed good reliability for healthy children and children with chronic medical conditions and their parents.
quality of life of families of children with CKD | 6 months
  The PedsQL FIM appears to be a useful tool for the assessment of family impact on children with ESRD

CONTACTS AND LOCATIONS:
Overall Officials: Amira M El Tohamy, Doctoral, Study Chair — Professor of pediatrics Faculty of Physical Therapy, Cairo University; Amira M Abd-Elmonem, Doctoral, Study Director — Assistant Professor of pediatrics Faculty of Physical Therapy, Cairo University; Rasha EE Galal, Doctoral, Study Director — Professor of pediatrics, Faculty of Medicine, Cairo University

REFERENCES:
- [Background] Abd El Basset Bakr AM, Hasaneen BM, AbdelRasoul Helal Bassiouni D. Assessment of Nutritional Status in Children With Chronic Kidney Disease Using Hand Grip Strength Tool. J Ren Nutr. 2018 Jul;28(4):265-269. doi: 10.1053/j.jrn.2017.12.007. Epub 2018 May 3. PMID 29731235
- [Background] Maher CA, Williams MT, Olds TS. The six-minute walk test for children with cerebral palsy. Int J Rehabil Res. 2008 Jun;31(2):185-8. doi: 10.1097/MRR.0b013e32830150f9. PMID 18467936
- [Background] Pathare N, Haskvitz EM, Selleck M. 6-Minute Walk Test Performance in Young Children who are Normal Weight and Overweight. Cardiopulm Phys Ther J. 2012 Dec;23(4):12-8. PMID 23304095
- [Background] Baek HS, Park KS, Ha IS, Kang HG, Cheong HI, Park YS, Lee JH, Cho HY, Cho MH. Impact of end-stage renal disease in children on their parents. Nephrology (Carlton). 2018 Aug;23(8):764-770. doi: 10.1111/nep.13083. PMID 28612957